CLINICAL TRIAL: NCT00262132
Title: Mycophenolate for Pulmonary Sarcoidosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CEL401; HR 11031
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: Mycophenolate

SUMMARY:
Corticosteroids are presently the drug of choice for the treatment of pulmonary sarcoidosis. However, corticosteroids are associated with many significant side effects. For this reason, it would be beneficial to find an alternative agent to corticosteroids for the treatment of pulmonary sarcoidosis. This study is an open label trial of mycophenolate for new onset pulmonary sarcoidosis. Patients are candidates for this study if they have biopsy proven pulmonary sarcoidosis and a vital capacity or FEV1 less than 80% of predicted. Patients must undergo bronchoscopy where not only is the diagnosis of pulmonary sarcoidosis required, but in addition, cells are obtained from bronchoalveolar lavage. If the patients are diagnosed with pulmonary sarcoidosis, they are placed on an initial dose of 500mg BID of mycophenolate for 1 week. If their blood counts are not affected on this dose and they have no significant symptoms that are thought to be drug related, then their dose is escalated to 1g BID for the remaining 9 weeks of the study (the total study drug therapy time is 10 weeks). The patients are followed with multiple study visits. At these visits blood tests are drawn to make sure that there are no significant side effects from mycophenolate. In addition, the patients have a history and physical performed to evaluate the clinical state of their sarcoidosis and to detect mycophenolate side effects. On completion of 10 weeks of mycophenolate therapy, the patients undergo a second bronchoscopy with bronchoalveolar lavage to obtain cells for analysis. The patients are evaluated with spirometry, measurements of shortness of breath (dyspnea), and a quality of life scale (SF36) at serial visits during their study. The primary endpoint of the study is improved, unchanged or worse FVC. It is hoped that this pilot study will suggest that mycophenolate is a reasonable treatment option for new onset pulmonary sarcoidosis.

ELIGIBILITY:
Inclusion criteria:

New acute pulmonary sarcoidosis defined as a FVC or FEV1 less than 80 percent of predicted plus symptoms of worsening dyspnea, cough, chest pain, or wheezing in patients without a prior history of pulmonary sarcoidosis. All such patients will also require bronchoscopy with transbronchial biopsy that demonstrates noncaseating granulomas of unknown cause. Such patients are usually treated for acute pulmonary sarcoidosis. The transbronchial biopsy specimens must have negative stains for mycobacteria and fungi.

> 18 years of age

Signing a written informed consent form.

Exclusion Criteria

1. Previous history of an adverse reaction to mycophenolate.
2. Current use of another immunosuppressive medication.
3. History of active hepatitis or another significant liver disease with the exception of proven or presumed sarcoidosis of the liver.
4. Previous history of skin cancer
5. Active peptic ulcer disease
6. Pregnant and/ or lactating female
7. Serum creatinine > 2.0 mg/dl
8. Serum bilirubin > 3.0 mg/dl
9. WBC < 4,000/cu mm3
10. Has demonstrated non-compliance in the past
11. Current alcohol or drug abuse
12. Evidence of significant sarcoidosis in extrapulmonary organs that requires therapy such that the mycophenolate doses could not be tapered if the pulmonary sarcoidosis was stable or improved.
13. History of previous severe digestive system disease
14. Patients taking azathioprine
15. Patients taking cholestyramine or other drugs that affect enterohepatic recirculation
16. Patients with Lesch-Nyhan or Kelley-Seegmiller syndrome
17. Patients be willing not to receive live vaccines during the study
18. Patients with phenylketonuria
19. Patients with elevated serum transaminases or total bilirubin at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Judson, MD, Principal Investigator — Medical University of South Carolina; Don C Rockey, MD, Study Chair — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States